CLINICAL TRIAL: NCT04102410
Title: Assessing Force-velocity Profile: an Innovative Approach to Optimize Cardiac Rehabilitation in Coronary Patients
Acronym: CITIUS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Saint Etienne (Other)
Collaborators: Jean Monnet University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 1708238; 2018-A01613-52 (Other: ANSM)
Record Dates: First submitted 2019-09-23; First posted 2019-09-25 (Actual); Last update posted 2022-06-03 (Actual); Status verified 2022-06

CONDITIONS: Acute Coronary Syndrome
Keywords: Cardiac rehabilitation; Physical activity; Force-velocity profile; Autonomic nervous system; Coronary artery disease
MeSH Terms: conditions — Acute Coronary Syndrome; Motor Activity; Coronary Artery Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): Patient with acute coronary syndrome will be included. They will have sprints, vertical jumps, questionary Short Form-12 (SF-12), activity actigraph and program composed of two 2 training strategies.
  Interventions: Other: Sprints; Other: Vertical jumps; Other: Questionary Short Form-12 (SF-12); Device: activity actigraph; Other: Program composed of two 2 training strategies
- Control group (Sham Comparator): Patient with acute coronary syndrome will be included. They will have sprints, vertical jumps, questionary Short Form-12 (SF-12), activity actigraph and program of usual practice.
  Interventions: Other: Sprints; Other: Vertical jumps; Other: Questionary Short Form-12 (SF-12); Device: activity actigraph; Other: Program of usual practice

INTERVENTIONS:
Other: Sprints — Two sprints of 8 seconds on a cycle ergometer will be performed for determine Force/Velocity Profile (FVP).
  Realized at inclusion and 2 months after.
Other: Vertical jumps — Two vertical jumps will be performed. Height of theses vertical jumps will be measured by application "My jump 2" to determine muscle power.
  Realized at inclusion and 2 months after.
Other: Questionary Short Form-12 (SF-12) — Questionary Short Form-12 (SF-12) will be performed to evaluate quality of life. It is composed of 12 questions.
  Realized at inclusion and 2 months after.
Device: activity actigraph — Activity actigraph will be wearing by patient during 7 consecutive days. It measures the level of physical activity and the sedentary lifestyle of patients.
  Realized at inclusion and 2 months after.
  Other Names: Wristlet connected
Other: Program composed of two 2 training strategies — Program composed of two 2 training strategies according to the initial Force/Velocity Profile (FVP) will be realized at the inclusion.
  There are :
  * Strategy "experimental-speed": speed training strategy for subjects with a force-speed profile (PFV) in favour of force
  * Strategy "experimental-force": force training strategy for subjects with a force-speed profile (PFV) in favour of speed.
  Arms: Experimental group
Other: Program of usual practice — Program composed of training in force and speed independently of the initial Force/Velocity Profile (FVP).
  Arms: Control group

SUMMARY:
Cardiac rehabilitation includes aerobic and anaerobic training adapted to cardiovascular pathology for which cardiac rehabilitation is prescribed. It is essential to adapt the content of these cardiac rehabilitation sessions to optimize aerobic and anaerobic performance and quality of life. Improvement of the first ventilatory threshold is one of the main objectives since it illustrates the adaptation of the patient to submaximal exercise, typical of everyday life.

The research laboratory "Autonomous Nervous System - Epidemiology, Physiology, Engineering, Health" (SPA-EPIS) has an international expertise in training optimization in top-athletes. He have shown the importance of the relationship between the power-force-velocity profile and athletes performances.

DETAILED DESCRIPTION:
In this sudy, each patient has a force and a velocity that can be optimized with training to achieve maximum power. This optimization can be evaluated through a force-velocity profile, measured from an only sprint on a cycloergometer.

The hypothesis that force-velocity profile could be used in cardiac rehabilitation in coronary patients to induce a force-velocity balance adapted through personalized sessions and regular medical follow-up.

This prospective, controlled, randomized and open label study will attempt to evaluate further the relevance of force or velocity training based on the initial force-velocity profile of coronary patients included in the cardiac rehabilitation program in the University Hospital of Saint-Etienne.

ELIGIBILITY:
Inclusion Criteria:

* Acute coronary syndrome treated within the last 6 months
* Medical revascularization (angioplasty ± stenting) or surgical (coronary artery bypass)
* During initial effort test: Maximum aerobic power≥ 60 watts for women and ≥ 80 watts for men
* Patient affiliated or beneficiary to social security
* Signed informed consent

Exclusion Criteria:

* Significant co-morbidities limited practice of physical activity
* Inability to submit to medical monitoring of the program
* Patient deprived of liberty or patient under guardianship
* Pregnant woman

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2019-09-30 (Actual); Primary Completion 2022-04-04 (Actual); Study Completion 2022-04-04 (Actual)

PRIMARY OUTCOMES:
volume of oxygen consumed (VO2) (in ml/min/kg) at the first ventilatory threshold (SV1) | Months: 0 and 2
  Change in VO2 (volume of oxygen in ml/min/kg) at the first ventilatory threshold (SV1) during a Cardio-Pulmonary Exercise Test (CPET).

SECONDARY OUTCOMES:
VO2 max (volume of oxygen maximum in ml/min/kg) | Months: 0 and 2
  Comparison VO2 max (volume of oxygen maximum in ml/min/kg) during a Cardio-Pulmonary Exercise Test (CPET).
Power at first ventilatory threshold (SV1) | Months: 0 and 2
  Comparison value of power at first ventilatory threshold (SV1) during a Cardio-Pulmonary Exercise Test (CPET).
Maximum aerobic power (in watt) | Months: 0 and 2
  Comparison maximum aerobic power (in watt) during a Cardio-Pulmonary Exercise Test (CPET).
Voluntary muscle power (in kg) during a static muscle testing on quadriceps | Months: 0 and 2
  Comparison voluntary muscle power (in kg) during a static muscle testing on quadriceps.
Voluntary muscle power (in kg) during a dynamic muscle testing on quadriceps | Months: 0 and 2
  Comparison voluntary muscle power (in kg) during a dynamic muscle testing on quadriceps.
Value of muscular endurance (in min) during a static muscle testing on quadriceps | Months: 0 and 2
  Comparison value of muscular endurance (in min) during a static muscle testing on quadriceps.
Value of muscular endurance (in min) during a dynamic muscle testing on quadriceps | Months: 0 and 2
  Comparison value of muscular endurance (in min) during a dynamic muscle testing on quadriceps.
Standard Deviation of the Normal R-R interval (SDNN) index | Months: 0 and 2
  Measured by holter electrocardiogram during 24 hours.
BaroReflex Sensitivity (BRS) (in ms/mmHg) | Months: 0 and 2
  Measured by baroreflex.
Physical activity (in Metabolic Equivalent of Task (MET)-min/week) | Month: 0
  Assessment of Physical activity (in Metabolic Equivalent of Task (MET)-min/week).
  Measured by activity actigraph.
Sedentary life (in hour/day) | Month: 0
  Assessment of Sedentary life (in hour/day). Measured by activity actigraph.
SF-12 questionnaire score | Months: 0 and 2
  The SF-12 is a self-questionnaire to assess the quality of life. This tool is an abbreviated version of the "Medical Outcomes Study Short-Form General Health Survey" (SF-36) contains only 12 items out of 36 with minimum score 0 (bad quality life) and maximum score at 100 (good quality life).

CONTACTS AND LOCATIONS:
Overall Officials: David HUPIN, MD, Principal Investigator — CHU SAINT-ETIENNE
Locations (1):
- Chu Saint-Etienne, Saint-Etienne, France

IPD SHARING:
Plan to Share IPD: No